CLINICAL TRIAL: NCT05584410
Title: Digitalization of the Care for Patients With Hip and Knee Osteoarthritis
Brief Title: Digitalization of Osteoarthritis Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Digitalization OA care
Record Dates: First submitted 2022-09-19; First posted 2022-10-18 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: physiotherapy; osteoarthritis; digital care
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis | interventions — Confidentiality; Blood Glucose Self-Monitoring

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- App-based model of care (Experimental): The app-based model of care includes at least one physical visit at the clinic. The majority of the treatment is provided by the app, containing five different sections:
  1) My information: specific information regarding osteoarthritis and generic lifestyle advice. 2 & 3) My exercise & My plan: individualized exercises where instructions are given through real-time video or pictures and written descriptions. The patient has access to a calendar and an overview of scheduled rehabilitation/exercises and care meetings. 4) My progress: weekly assessment of pain + every six-month with valid patient reported outcome measures and test of function. 5) My messages (asynchronous chat with the responsible physiotherapist). The app sends automatic and daily reminders and / or motivational notifications.
  Interventions: Other: Patient information; Other: Smart phone application based exercises; Other: Self-monitoring; Behavioral: Motivational notifications
- Web-based model of care (Active Comparator): The patient will get access to information about osteoarthritis and generic osteoarthritis exercises program from a web-based platform Individualization of the training can be done by the responsible physiotherapist informing about changes in the training via the message function and / or during physical follow-up visits. An individualized rehabilitation program can be given to the patient, via the platform or at a physical visit at the clinic, in form of a document with pictures and descriptive information. As long as the patient is under treatment (approximately three months), he/she can contact their responsible physiotherapist by sending a message from the platform.
  Interventions: Other: Patient information; Other: Web based exercises; Other: Home based rehabilitation
- Standard care (Active Comparator): Patients who are randomized to standard care receive osteoarthritis specific information at three different group meetings (physical or digital) led by a physiotherapist, an occupational therapist and / or dietitian (each rehab clinic makes its own arrangement). After the theory sessions, the patient is booked for another physical visit to the responsible physiotherapist where an individual training program is tested. The patient is then offered to regularly exercise at the clinic, individually or in a group under supervision from a physiotherapist.
  Interventions: Other: Patient information; Other: Group based information; Other: Supervised rehabilitation; Other: Home based rehabilitation

INTERVENTIONS:
Other: Patient information — Patient education according to national guidelines, with information about e.g. disease progression, symptoms, treatment, exercise, self-care techniques and dietary information
Other: Smart phone application based exercises — Individually based exercise programs individualized exercises where instructions are given through real-time video or pictures in combination with written descriptions.
  Arms: App-based model of care
Other: Web based exercises — Generic osteoarthritis exercise, including about 20 different exercises, provided by real-time videos and written description
  Arms: Web-based model of care
Other: Group based information — Osteoarthritis specific information at three different group meeting (physical or digital) led by a physiotherapist, an occupational therapist and / or dietitian (each rehab clinic makes its own arrangement).
  Arms: Standard care
Other: Supervised rehabilitation — The patient is offered to regularly exercise at the clinic, individually or in a group under supervision from a physiotherapist.
  Arms: Standard care
Other: Self-monitoring — Patients will be followed by validated questionnaires and function tests (30 sec Chair-to-stand test) every six months until three years after the start of treatment. The patients will get a report of the results and a research coordinator will contact the patients if their symptoms/function has worsen and discuss further treatment
  Arms: App-based model of care
Behavioral: Motivational notifications — Automatic and daily reminders and / or motivational notifications
  Arms: App-based model of care
Other: Home based rehabilitation — Individualized exercises that the patient performs on their own, i.e. at home or at a gym.
  Arms: Standard care; Web-based model of care

SUMMARY:
The overall aim of this study is to compare three different care models for patients with hip- and knee osteoarthritis. The primary aim is to evaluate whether an app-based care model is more beneficial for improving function in daily life than a web-based care model and standard care for patients with hip and / or knee osteoarthritis

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate whether an app-based care model is more beneficial for improving function in daily life than a web-based care model and standard care for patients with hip and / or knee osteoarthritis. The secondary aims are to evaluate how 1) patient-related outcome measures regarding the ability of the patient to "forget" about their problematic joint after treatment, quality of life, pain-related self-efficacy, and level of physical activity and 2) care consumption, cost-effectiveness, and carbon footprint differ between the three care models in a short-term (three months) and long-term perspective (one and three years respectively). Further aims are to evaluate how patient experience of the benefits provided by the two digital care models differs, how patient experience with respect to work alliance differs between the three care models, describe the adherence to using the app in the app-based care model and to describe what patient characteristics are associated with clinically meaningful improvements in function in daily life among patients recieving app-based care. The primary hypothesis is that patients who are randomized to an app-based care model will improve significantly more in terms of function in daily life from baseline to one year compared with patients who are randomized to a web-based model and usual care. The secondary hypothesis is that patients randomized to the app-based care model change equivalently from baseline to one year in terms of patient-reported measures, but that the app-based care model is more cost-effective compared with the other two care models at one and three years, respectively.

ELIGIBILITY:
Inclusion Criteria:

The participant:

* has given their written consent to participate in the study
* has been referred to the orthopaedic clinic at Sahlgrenska University Hospital /Mölndal for primary hip- and or knee osteoarthritis
* has a positive attitude in using digital tools
* has access to a smart phone / tablet
* has been assessed not to be in need of hip or knee surgery trough triage based on a patient reported outcome (the Osteoarthritis Guidelines Instrument)

Exclusion Criteria:

Patients:

* with secondary osteoarthritis (due to osteonecrosis)
* referred to a specific orthopaedic surgeon
* with impaired mental ability, reluctance or language difficulties that make it difficult to understand the meaning of participating in the study
* who undergo treatment, have disability or illness that according to the research group can affect the treatment or the study result

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Hip dysfunction/Knee Osteoarthritis Outcome Score (HOOS/KOOS) subscale Function in daily living (ADL) | baseline to 12 months after inclusion
  The KOOS/HOOS questionnaires were developed as instruments to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale (scoring instructions are available in a separate document).
Hip dysfunction/Knee Osteoarthritis Outcome Score (HOOS/KOOS) subscale Function in daily living (ADL) | baseline to 36 months after inclusion
  The KOOS/HOOS questionnaires were developed as instruments to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale (scoring instructions are available in a separate document).

SECONDARY OUTCOMES:
Hip dysfunction/Knee Osteoarthritis Outcome Score (HOOS/KOOS) subscale pain, symptoms, function in sport and recreation, and knee/hip related quality of life | baseline
  The KOOS/HOOS questionnaires were developed as instruments to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale (scoring instructions are available in a separate document).
Hip dysfunction/Knee Osteoarthritis Outcome Score (HOOS/KOOS) subscale pain, symptoms, function in sport and recreation, and knee/hip related quality of life | 3 months after inclusion
  The KOOS/HOOS questionnaires were developed as instruments to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale (scoring instructions are available in a separate document)
Hip dysfunction/Knee Osteoarthritis Outcome Score (HOOS/KOOS) subscale pain, symptoms, function in sport and recreation, and knee/hip related quality of life | 12 months after inclusion
  The KOOS/HOOS questionnaires were developed as instruments to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale (scoring instructions are available in a separate document).
Hip dysfunction/Knee Osteoarthritis Outcome Score (HOOS/KOOS) subscale pain, symptoms, function in sport and recreation, and knee/hip related quality of life | 36 months after inclusion
  The KOOS/HOOS questionnaires were developed as instruments to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale (scoring instructions are available in a separate document).
The Forgotten joint score (hip/knee) (FJS) | baseline
  A questionnaire that was developed to find subtle differences between patients who grade their hip / knee as "very good" and "excellent". The score is graded from 0 to 100, where a higher score is better.
The Forgotten joint score (hip/knee) (FJS) | 3 months after inclusion
  A questionnaire that was developed to find subtle differences between patients who grade their hip / knee as "very good" and "excellent". The score is graded from 0 to 100, where a higher score is better.
The Forgotten joint score (hip/knee) (FJS) | 12 months after inclusion
  A questionnaire that was developed to find subtle differences between patients who grade their hip / knee as "very good" and "excellent". The score is graded from 0 to 100, where a higher score is better.
The Forgotten joint score (hip/knee) (FJS) | 36 months after inclusion
  A questionnaire that was developed to find subtle differences between patients who grade their hip / knee as "very good" and "excellent". The score is graded from 0 to 100, where a higher score is better.
Swedish National Board of Health and Welfare questions about physical activity | baseline
  Questions intended for use in clinical health care to identify people that are insufficiently physically active. The respondents report their total time, in minutes, of moderate and vigorous physical activity, respectively, during a normal week on a categorical scale from a) 0-30 minutes, up to g) >300 minutes.
Swedish National Board of Health and Welfare questions about physical activity | 3 months after inclusion
  Questions intended for use in clinical health care to identify people that are insufficiently physically active. The respondents report their total time, in minutes, of moderate and vigorous physical activity, respectively, during a normal week on a categorical scale from a) 0-30 minutes, up to g) >300 minutes.
Swedish National Board of Health and Welfare questions about physical activity | 12 months after inclusion
  Questions intended for use in clinical health care to identify people that are insufficiently physically active. The respondents report their total time, in minutes, of moderate and vigorous physical activity, respectively, during a normal week on a categorical scale from a) 0-30 minutes, up to g) >300 minutes.
Swedish National Board of Health and Welfare questions about physical activity | 36 months after inclusion
  Questions intended for use in clinical health care to identify people that are insufficiently physically active. The respondents report their total time, in minutes, of moderate and vigorous physical activity, respectively, during a normal week on a categorical scale from a) 0-30 minutes, up to g) >300 minutes.
Heath-related quality of life - EuroQol (EQ5-D) | baseline
  Measure of health-related quality of life and consists of 5 items. General health is measured using a visual analog scale (0 to 100) with 100 being the best possible health state.
Heath-related quality of life - EuroQol (EQ5-D) | 3 months after inclusion
  Measure of health-related quality of life and consists of 5 items. General health is measured using a visual analog scale (0 to 100) with 100 being the best possible health state.
Heath-related quality of life - EuroQol (EQ5-D) | 12 months after inclusion
  Measure of health-related quality of life and consists of 5 items. General health is measured using a visual analog scale (0 to 100) with 100 being the best possible health state.
Heath-related quality of life - EuroQol (EQ5-D) | 36 months after inclusion
  Measure of health-related quality of life and consists of 5 items. General health is measured using a visual analog scale (0 to 100) with 100 being the best possible health state.
Medtech20 | 3 months after inclusion
  A standardized tool measuring how medical devices affect people's sense of security, integrity, social participation and convenience. Each item is rated on a seven graded Likert-scale from, 0 = "disagree" to 6 = "completely agree". Each item also has a "Not applicable" response option. A higher score indicates a better effect of the medical device.
Working Alliance Inventory-Short Revised | 3 months after inclusion
  A recently refined measure of the therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. The questionnaire is validated, has acceptable reliability and includes 12 items. The patient rates each item on a seven graded Likert-scale from 1 = "not at all" to 7 = "completely". A higher score indicates a better therapeutic alliance.
Pain Self-Efficacy Scale - 2 item | baseline
  The Pain Self-Efficacy Questionnaire (PSEQ) is an established 10-item measure of pain self-efficacy that is widely used in clinical and research settings. In the present study a short form of the original questionnaire will be used. The two items are graded from 0 = not at all certain to 6 = very certain.
Pain Self-Efficacy Scale - 2 item | 3 months after inclusion
  The Pain Self-Efficacy Questionnaire (PSEQ) is an established 10-item measure of pain self-efficacy that is widely used in clinical and research settings. In the present study a short form of the original questionnaire will be used. The two items are graded from 0 = not at all certain to 6 = very certain.
Pain Self-Efficacy Scale - 2 item | 12 months after inclusion
  The Pain Self-Efficacy Questionnaire (PSEQ) is an established 10-item measure of pain self-efficacy that is widely used in clinical and research settings. In the present study a short form of the original questionnaire will be used. The two items are graded from 0 = not at all certain to 6 = very certain.
Pain Self-Efficacy Scale - 2 item | 36 months after inclusion
  The Pain Self-Efficacy Questionnaire (PSEQ) is an established 10-item measure of pain self-efficacy that is widely used in clinical and research settings. In the present study a short form of the original questionnaire will be used. The two items are graded from 0 = not at all certain to 6 = very certain.
Cost Effectiveness | 3 months after inclusion
  Indirect and direct health care costs. Total costs, costs per patient and per visit. Loss of income will be reported as number of days of abscence due to illness.
Cost Effectiveness | 12 months after inclusion
  Indirect and direct health care costs. Total costs, costs per patient and per visit. Loss of income will be reported as number of days of abscence due to illness.
Cost Effectiveness | 36 months after inclusion
  Indirect and direct health care costs. Total costs, costs per patient and per visit. Loss of income will be reported as number of days of abscence due to illness.
Assessment of carbon dioxide (CO2) equivalent emissions in kg - travelling | Baseline
  Travelling to/from health care visits based on travel data reported in a questionnaire
Assessment of CO2 equivalent emissions in kg - electronical devices | 3 months after inclusion
  Use of electronical devices in a lifecycle perspective based on user data from app

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kilhamn, PhD, Principal Investigator — Research, Education, Development & Innovation, Primary Health Care, Region Västra Götaland, Sweden
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Time Frame: Data will become available after publication of results
Access Criteria: Analyses and additional data are available upon request